CLINICAL TRIAL: NCT02294955
Title: Catheter Ablation Compared With Pharmacological Therapy for Atrial Fibrillation - a Randomized Multicentre Study Comparing Atrial Fibrillation Ablation Strategy With Optimized Conventional Pharmacological Strategy After 12 Months Follow-up.
Brief Title: Catheter Ablation Compared With Pharmacological Therapy for Atrial Fibrillation (CAPTAF Trial)
Acronym: CAPTAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Carina Blomstrom Lundqvist, Professor, Senior consultant, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-001384-11
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation; Quality of Life
Keywords: catheter ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; Sotalol; Flecainide; Propafenone; Disopyramide; Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheterablation (Active Comparator): Pulmonary vein isolation with Cryo-energy using a Arctic Front™ Cardiac CryoAblation Catheter or an irrigated radiofrequency ablation catheter, with an optional roof line.
  Interventions: Drug: Amiodarone; Drug: Sotalol; Drug: Flecainide; Drug: Propafenone; Drug: Disopyramide; Drug: Dronedarone
- Antiarrhythmic drug Class IC or III. (Active Comparator): Serial testing of oral antiarrhythmic drugs; amiodarone 600 mg once daily 7-10 days, then 100-200 mg once daily; sotalol: 80-160 mg twice daily; flecainide 100 to 150 mg twice daily or entire dose as slow-release formula once daily; propafenone 300 mg twice daily; disopyramide 250-375mg twice daily, or dronedarone 400 mg twice Daily.
  Interventions: Device: Catheterablation

INTERVENTIONS:
Device: Catheterablation — Pulmonary vein isolation using either Arctic Front™ Cardiac CryoAblation or irrigated radiofrequency catheter ablation. A linear lesion, a left atrial roof line, is optional for patients with AF recurrence after a first procedure or primarily for patients with persistent AF.
  Arms: Antiarrhythmic drug Class IC or III.
Drug: Amiodarone — Dosage orally 600 mg once daily for 7-10 days, and 100-200 mg once daily thereafter.
  Other Names: Cordarone®
  Arms: Catheterablation
Drug: Sotalol — Dosage orally 80-160 mg twice daily
  Other Names: Sotalol®
  Arms: Catheterablation
Drug: Flecainide — Dosage orally 100 to 150 mg twice daily or the entire dose as slow-release formula once daily
  Other Names: Tambocor®
  Arms: Catheterablation
Drug: Propafenone — Dosage orally 300 mg twice daily
  Other Names: Rythmol®
  Arms: Catheterablation
Drug: Disopyramide — Dosage orally 250-375 mg twice Daily
  Other Names: Norpace®
  Arms: Catheterablation
Drug: Dronedarone — Dosage orally 400 mg twice daily
  Other Names: Multaq®
  Arms: Catheterablation

SUMMARY:
The objective is to compare the efficacy of 2 treatment strategies, catheter ablation of atrial fibrillation versus optimized pharmacological therapy, in patients with symptomatic atrial fibrillation.

It is a randomized, prospective, controlled, open-label multicentre, parallel-group study including 116 patients. Inclusion criteria are patients aged 30-70 years with symptoms related to atrial fibrillation and who have failed or been intolerant to at least one anti-arrhythmic drug, with at least one atrial fibrillation episode documented on ECG during the previous 12 months and at least one symptomatic episode during the previous 2 months or at least 2 symptomatic episodes of persistent AF in the previous 12 months.

Main exclusion criteria are patients who have tested 2 or more anti-arrhythmic drugs for rhythm control, uncontrolled hypertension, valvular disease requiring anticoagulation, planned valve surgery within 2 years, contraindication to treatment with anticoagulants, heart failure, left atrial diameter > 60 mm, unstable angina or acute myocardial infarction within the last 3 months, cardiac revascularization procedure within the last 6 months, prior cardiac surgery or planned cardiac corrective surgery within 1 year, prior AF ablation procedure.

The primary endpoint is general health-related quality of life at 12 months follow-up. The main secondary endpoints are morbidity and mortality as composite outcome, cardiovascular hospitalization, symptoms, heart failure, left atrial and ventricular function and diameters, exercise capacity, health care economics, rhythm, atrial fibrillation burden, successful versus failed treatment, safety and "cross-overs" over time.

Patients will receive a cardiac monitor, implanted subcutaneously, which will monitor the heart rhythm during a two month "Run-in" period, for the definition of the basic atrial fibrillation burden. Patients will be randomly assigned to an antiarrhythmic drug (for rhythm or rate control) or to left atrial catheter ablation. Evaluation of outcome is at 12, 24, 36 and 48 months of follow-up, while health economy will be evaluated at 24 and 48 months of follow-up.. In case of documented disease progression or unacceptable toxicity, subjects will be switched to the alternative regimen. The main statistical analysis of the primary endpoint will be based on the intention-to-treat population. The trial duration is 48 months.

DETAILED DESCRIPTION:
It is a randomized, open-label, multi-centre trial in which patients with symptomatic paroxysmal or persistent atrial fibrillation will be randomized to treatment with either catheter ablation for pulmonary vein isolation or optimized conventional pharmacological therapy. Patients will receive an implantable cardiac monitor, Reveal XT, implanted subcutaneously, before a two month "Run-in" period from which the basic atrial fibrillation burden will be defined, which will provide an objective basis to assess the AF burden for 3 years.

After initiation of randomized therapy, patients will be followed at 3, 6, 9, 12, 18, 24, 30, 36 and 48 months. In case of intolerable symptomatic atrial fibrillation despite allocated treatment, subjects will be switched to the alternative regimen, on patient's request.

The ablation will consist of pulmonary vein isolation for both paroxysmal and persistent atrial fibrillation. A linear lesion at the left atrial roof is optional for patients with recurrence after a first procedure or primarily for patients with persistent atrial fibrillation only. A second ablation procedure may be undertaken at earliest 3 months after the first procedure, if symptoms persists or recurs. Epicardial off-pump ablation may be offered after failed attempts of transvenous catheter ablation at earliest 3 months after latest procedure. If the second transvenous ablation procedure fails, patients may be offered i) a third transvenous ablation procedure or ii) an epicardial off-pump procedure. In case the patient declines a third intervention despite recurrence, the patient should continue on the same anti-arrhythmic drugs. If new previously untested drugs are prescribed, the patient will be defined as a change of treatment (and failed ablation). Ablation may be performed using radiofrequency energy with irrigated tip or with cryo-energy using the Arctic Front™ Cardiac CryoAblation Catheter. A complete pulmonary vein isolation will be defined by documenting PV entrance block in each vein using a circular mapping catheter.

Anti-arrhythmic drugs remaining to be tested for rate and rhythm control may include previously tested tolerable antiarrhythmic drugs if dosages were inadequate. Optimized anti-arrhythmic drug therapy includes testing of all available anti-arrhythmic drugs at adequate dosages, including amiodarone 600 mg once daily for 7-10 days, and 100-200 mg once daily thereafter; sotalol: 80-160 mg twice daily; flecainide 100 to 150 mg twice daily or the entire dose as slow-release formula once daily; propafenone 300 mg twice daily; and disopyramide 250-375mg twice daily, and potentially new antiarrhythmic drugs commercially available during the study period.

A monitor will verify that data recorded on the procedure forms are correct through quarterly communication, review of catheterization reports and medical records. In accordance with applicable regulations a monitor (study nurse from Uppsala) will contact the site prior to the start of the study to review with the site staff protocol, study requirements and their responsibilities to satisfy study requirements, if needed. When reviewing data collection procedures the discussion will also include identification, agreement and documentation of data items for which the case record forms (CRF), patient files (paper or database), tracings of investigations, and questionnaires, will serve a source document. The investigator and the head of the medical institution agrees should allow the monitor direct access to all relevant documents whenever needed and in an event of an audit. To ensure compliance the monitor may conduct a quality assurance audit, which can occur at any time during or after completion of the study.

The Biometrics section at Uppsala Clinical Research Centre is responsible for the Data Management. All data will be recorded in the CRFs and entered via eCRF directly into a web based data capturing system except for electronically available data that will be loaded directly into the study database. Each investigational site will have authorized site personnel responsible for entering the data, as well as for changing and correcting the data according to instructions provided by Uppsala Clinical Research Centre (UCR) and the coordinating centre. All changes will be tracked by an audit trail. The site specific investigator will sign the eCRF electronically when the data have been reviewed and edited, and Source Data Verification has been performed.

The Database Closure will be performed in three steps, the first one when all data from the first 12 months are entered, the second one when all data from the 24 months period are entered and the third when the complete study period of 48 months are entered. All datasets used for the 12- and 24 months analyses will be locked separately. Procedures: When all data are entered into the database and all queries solved, the Database Closure procedures will start.

Complications are defined as acute if occurring within 1 week after initialized therapy, and late if occurring one week after initialized therapy. All "Serious adverse events" should be documented on the "Adverse events Form" AND "Serious adverse events Form". All " Adverse events" should be documented in the "Adverse events Form". All events which are part of performing a catheterization procedure will be reported. All serious unanticipated events whether or not they are considered to be related to the procedure but which have some association with the catheterization either by timing or physiology, will be reported. Other bleedings than major bleeding events should be reported as minor bleeds. All events related to pharmacological therapy will be reported.

Procedural complications are defined as those arising during or within 1 month of the procedure, including death, major bleeding, vascular injury, cerebrovascular accident, myocardial infarction, pericardial effusion with or without tamponade, venous or systemic embolism, phrenic nerve paralysis, and heart block. Events occurring later than 1 month after the procedure and defined as related to the procedure are pulmonary vein stenosis, tamponade, retroperitoneal haematoma, and atrio-esophageal fistula (see below).

Relation to Device Procedure or drug, Intensity, Outcome and Actions taken will be described according to international regulations.

Statistical methods. All continuous variables will be presented per treatment group using descriptive statistics by mean, SD, max and min values, in addition medians, 25th and 75th percentiles will be presented when suitable.

The analysis of mean change in the primary endpoint will be two-sided and performed as an unpaired t-test at 5% significance level. The difference between the treatment groups with corresponding two-sided 95% confidence interval based on a normal approximation will be presented. The continuous secondary endpoints will be analyzed in the same way as the primary endpoint, but the results will be interpreted descriptively. Kaplan-Meier estimates and log-rank test will be used to determine the occurrence of the secondary endpoints over time. All categorical secondary endpoints will be compared between treatment groups with frequency tables and Fisher's Exact Test including 95% confidence intervals where possible. Adverse Events will be summarized per treatment group by body system/system organ class, preferred terms, intensity, seriousness and relationship. Laboratory data for efficacy will be presented in mean change tables.

The null hypothesis (H0) is that the difference in the mean change from baseline to 12 months after baseline in General Health between the two treatments is zero;- mean change for the treatment group catheter ablation (μ 1) and - mean change for the treatment group optimized conventional pharmacological therapy (μ 2) Safety - All randomized patients will be included in the safety analysis. Only observed observations are used in the safety analysis.

Intention to treat (ITT) - All randomized patients. The main analysis will be performed on the ITT-population.

Per protocol (PP) - All randomized patients completing the study treatment period of 12 months without any major protocol violation (for example ineligibility, early withdrawals, poor compliance).

A subgroup analysis will determine whether sinus rhythm obtained by AF ablation is superior to sinus rhythm obtained by pharmacological therapy for rate and/or rhythm control. In addition a comparison will be done between patients with sinus rhythm and patients with atrial fibrillation irrespective of allocated therapy. Both analyses will be performed with regard to quality of life, morbidity (composite, see secondary endpoint 1), cardiovascular hospitalizations, exercise/ physical capacity, safety, and health economy at 12 and 24 months.

All continuous variables will be presented per treatment group using descriptive statistics by mean, standard deviation, max and min values, in addition medians, 25th and 75th percentiles will be presented when suitable. The analysis of mean change in the primary endpoint will be two-sided and performed as an unpaired t-test at 5% significance level. The difference between the treatment groups with corresponding two-sided 95% confidence interval based on a normal approximation will be presented.

The continuous secondary endpoints will be analyzed in the same way as the primary endpoint, but the results will be interpreted descriptively.

Kaplan-Meier estimates and log-rank test will be used to determine the occurrence of the secondary endpoints over time. All categorical secondary endpoints will be compared between treatment groups with frequency tables and Fisher's Exact Test including 95% confidence intervals where possible. Adverse Events will be summarized per treatment group by body system/system organ class, preferred terms, intensity, seriousness and relationship.

Sample size considerations: The primary endpoint is the change in General Health from baseline to 12 months after baseline. Based on previous studies it is assumed that the variable is normally distributed with a standard deviation for the change in General Health of 20 units and an expected difference between groups of at least 10.5 units. To detect a difference of 10.5 units in General Health (corresponding to an improvement of 15%, assuming a mean General Health of 70 units in the conventional pharmacological therapy group) with a power of 80% and a type I error of 5% (two-sided alternative), a sample size of approximately 58 subjects in each treatment group is required, i.e. a total number of 116 patients. Another 20 patients are added to ensure calculated number of patients for analysis at 12 months. The power to detect a difference of 10.5 for 136 (116+20) and 140 (the minimum expected total number) patients is 85% and 86%, respectively.

A 1:1 block randomization will be used within each centre, stratifying patients between paroxysmal and persistent AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptoms related to atrial fibrillation (AF), who have failed or been intolerant to at least one drug used for either rate or rhythm control (Vaughan Williams class I, II, or III anti-arrhythmic drug) thus excluding digitalis and Calcium channel inhibitors.
2. The first diagnosis of AF must have been first noted more than 6 months prior to consideration.
3. At least one AF episode documented on 12-lead ECG or 2-channel telemetry/ Holter recording during the previous 12 months.
4. Paroxysmal AF (AF is self-terminating within 7 days of recognized onset) with occurrence of at least one symptomatic episodes (patient history) in the previous 2 months that merits non-pharmacological intervention (see classification), or
5. Persistent AF (AF is not self-terminating within 7 days or is terminated electrically or pharmacologically) with occurrence of at least 2 symptomatic episodes of AF in the previous 12 months, necessitating pharmacological or electrical cardioversions (CV), on or off antiarrhythmic drugs that merits non-pharmacological intervention. Upon cardioversion, it must be documented that sinus rhythm can be maintained for at least 1 hour, to distinguish from permanent AF.

Exclusion Criteria:

1. Patients who have tested 2 or more anti-arrhythmic drugs for rhythm control at highest tolerable dosages (Vaughan Williams class I or III anti-arrhythmic drug; flecainide, propafenone, disopyramide, sotalol or amiodarone).
2. AF secondary to a transient or correctable abnormality including electrolyte imbalance, trauma, recent surgery, infection, toxic ingestion, and uncontrolled thyroid disease.
3. Atrial fibrillation episodes triggered by another uniform supraventricular tachycardia.
4. Untreated or uncontrolled hypertension
5. Valvular disease requiring chronic anticoagulation or planned valve surgery within 2 years.
6. Contraindication to treatment with Warfarin or other anticoagulants.
7. Heart failure with New York Heart Association (NYHA ) class III or IV or left ventricular ejection fraction (LVEF) < 35 %, which is not secondary to AF with inadequate rate control, according to the judgement of the investigator.
8. Left atrial diameter > 60 mm.
9. Unstable angina or acute myocardial infarction within last 3 months.
10. Cardiac revascularization procedure within last 6 months.
11. Prior cardiac surgery or planned cardiac corrective surgery within 1 year.
12. Prior AF ablation procedure
13. Implantable cardioverter-defibrillator, biventricular pacing device, Dual chamber- and single chamber -pacemaker if needed for ventricular pacing, as well as Atrioventricular (AV) block II-III and sustained ventricular tachyarrhythmias.
14. Patients with intra-atrial thrombus, tumor, or another abnormality in whom transseptal catheterization or appropriate vascular access is precluded.
15. Renal failure requiring dialysis or abnormalities of liver function tests
16. Participant in investigational clinical or device trial.
17. Pregnant women.
18. Unwilling or unable to give informed consent or inaccessible for follow-up. Specify if implantable cardiac monitor (ICM) was not accepted by the patient to be implanted.
19. Psychological problem that might limit compliance.
20. Active abuse of alcohol or other substance which may be causative of AF and/or might affect compliance.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-05; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
quality of life | 12 months
  General Health related Quality of Life; Short Form (SF) 36

SECONDARY OUTCOMES:
atrial fibrillation burden | 12, 24, 36 and 48 months
  Total time spent in and number of episodes of atrial fibrillation, Frequency of symptomatic respectively asymptomatic episodes of AF assessed by implantable event recorder.
Composite of morbidity | 12, 24, 36 and 48 months
  Stroke, systemic embolic events, transient ischemic attack (TIA), major bleeding, cardiovascular hospitalizations, pacemaker implantation, all cause Death.
Hospitalization | 12, 24, 36 and 48 months
  Total number of hospitalization days and time to first event of hospitalization days due to cardiovascular reasons and atrial fibrillation
Quality of Life | 12, 24, 36 and 48 months
  Quality of Life by SF-36, all domains and time-points; symptom severity score (SSQ); European Heart Rhythm Association (EHRA) Symptom Classification.
Health care use and economy | 24 and 48 months
  EuroQoL (EQ) 5D, a standardised instrument for measure of health outcome, COSTs for hospitalization and outpatient visits related to and not related to AF, treatment costs, and including corrections for background variables regarding social economic status.
Success of treatment | 12 and 48 months
  Baseline predictors for symptom-based response (symptom success) and rhythm-based response.
Physical capacity | 12, 24, 36 and 48 months
  Exercise/Physical capacity and % of predicted max. as well as duration
Atrial area and function | 12, 24, 36 and 48 months
  Left atrial area and function, Right atrial area and function (from Echocardiography and corrected for body surface area.
Adverse events | 12, 24, 36 and 48 months
  Incidence, intensity and relationship of Adverse Events
Recurrence of episodes of AF lasting at least one minute. | 12, 24, 36 and 48 months
  After four weeks stabilization period, obtained from the implantable cardiac monitor and 24 hour Holter recordings and extra visits related to AF.
Success/failure of treatment. | 12, 24, 36, 48 months
  Success/failure (yes/no) with regard to symptoms and rhythm.

OTHER OUTCOMES:
Covariate adjusted primary endpoint | 12, 24, 36 and 48 months
  Analysis of primary endpoint using following covariates at baseline: age, sex, background variables regarding social economic status, BMI, paroxysmal or persistent AF type I or II, coronary artery disease, hypertension, diabetes, congestive heart failure, failure of an antiarrhythmic drug class I or III prior to randomization, present medication and duration of AF
Recurrence of episodes of AF lasting at least one minute | 12, 24, 36 and 48 months
  Recurrence of episodes of AF lasting at least one minute (after four weeks stabilization period), obtained from the ICM continuously and 24 hour Holter recordings and extra visits related to AF cardioversion).
Baseline predictors for symptom-based response and rhythm-based response. | 12, 24, 36 and 48 months
  Logistic multiple regression analysis to identify baseline predictors for symptom-based response (symptom success) and rhythm-based response (rhythm success if absence of AF episodes duration > 1 minute after last therapy), respectively (yes/no) by treatment Group.

CONTACTS AND LOCATIONS:
Overall Officials: Carina M Blomström Lundqvist, Professor, Principal Investigator — Department of Cardiology, University Hospital in Uppsala
Locations (1):
- Carina Blomström Lundqvist, Uppsala, Sweden